CLINICAL TRIAL: NCT05897632
Title: CARE-CP (Testing a Cardiovascular Ambulatory Rapid Evaluation for Patients With Chest Pain )
Brief Title: CARE-CP (Testing a Cardiovascular Ambulatory Rapid Evaluation for Patients With Chest Pain)
Acronym: CARE-CP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00092604
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-04

CONDITIONS: Chest Pain
Keywords: Acute Coronary Syndrome; Cardiovascular Diseases
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Patients will be randomized with equal probability (1:1) to the outpatient arm or the hospitalization arms using permuted block randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatient Evaluation (Other): Patients randomized to this arm are discharged and receive outpatient evaluation, or cardiovascular ambulatory rapid evaluation (CARE), focused on medical management for cardiovascular risk factors (e.g. hypertension) within 72 hours of Emergency Department discharge.
  Interventions: Behavioral: Outpatient Evaluation
- Hospitalization Evaluation (Other): Patients randomized to this arm receive evaluation for their symptoms in a hospital ward, observation unit, or emergency department boarding.
  Interventions: Behavioral: Hospitalization Evaluation

INTERVENTIONS:
Behavioral: Outpatient Evaluation — Subjects will receive an outpatient evaluation within 72 of being discharged from the ED.
  Other Names: CARE-CP (Cardiovascular Ambulatory Rapid Evaluation)
  Arms: Outpatient Evaluation
Behavioral: Hospitalization Evaluation — Patients randomized to this arm receive evaluation for their symptoms in a hospital ward, observation unit, or emergency department boarding.
  Arms: Hospitalization Evaluation

SUMMARY:
The goal of this study is to determine if rapid outpatient evaluation vs hospitalization management is the best strategy (based on patient-centered measures and safe, equitable, and efficient resource use) for evaluating patients with acute chest pain who are at moderate risk for acute coronary syndrome (ACS). Patients will be randomized in the Emergency Department to either an outpatient evaluation (CARE-CP) or hospitalization evaluation for their symptoms.

DETAILED DESCRIPTION:
Current care patterns for the 7 million patients visiting Emergency Departments (EDs) in the United States with chest pain are heterogeneous and not sustainable from a healthcare quality or economic perspective. Chest pain is the second most common cause of ED visits and the most common reason for short-stay hospitalizations. During these hospitalizations patients undergo in-depth evaluations (stress testing, computed tomography coronary angiography, or invasive angiography), but ultimately <10% are diagnosed with acute coronary syndrome (ACS). These evaluations cost $3 billion annually and strain health system resources without clear evidence of improved health outcomes or patient experience. The preliminary data suggest that moderate risk patients (35% of patients with chest pain) can be safely managed as outpatients using a cardiovascular ambulatory rapid evaluation (CARE-CP) strategy as an alternative to hospitalization. In the CARE-CP strategy, patients are discharged from the ED and receive outpatient clinic follow-up within 72 hours focused on medical management for cardiovascular risk factors (e.g., hypertension, diabetes) and determining whether further cardiac testing is needed. This strategy aims to enhance patient-centered outcomes while safely and equitably decreasing hospital resource utilization. However, equipoise exists between outpatient and hospitalization strategies for moderate risk patients. There is a paucity of prospective data evaluating the efficacy and patient-centeredness of outpatient chest pain evaluation strategies in moderate risk patients. Thus, it is unclear whether use of an outpatient chest pain management strategy (CARE-CP) will safely reduce healthcare utilization and be preferred by patients compared to a traditional hospitalization strategy. To address this key evidence gap, the study proposes the first prospective multisite randomized trial testing outpatient vs hospitalization strategies in moderate risk patients. The research teams will randomize 502 patients 1:1 to the CARE-CP or hospitalization management arms at three ED sites with a history of high recruitment rates and productive collaborations in cardiovascular clinical trials. The primary outcome will be hospital-free days (HFD) over a 30-day period. This novel trial addresses a key evidence gap by providing guidance on how best to evaluate moderate risk ED patients with acute chest pain. Without this guidance care patterns are likely to remain heterogeneous, inefficient, non-patient-centered, and unguided by the highest level of evidence. We hypothesize that data from this trial will support widespread implementation of a CARE-CP strategy, which could improve the quality and value of care for millions of patients in the U.S. and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21 years old
* Chest pain or Symptoms of acute coronary syndrome (ACS)
* Moderate risk of ACS (all of the below)
* Hear Score 4-6
* Non-Ischemic electrocardiogram (ECG)
* Two Troponin measures < Sex-Specific Upper Reference Limit

  * Women <15 pg/ml
  * Men <20 pg/ml
* No prior coronary artery disease (CAD)

  * No Prior Myocardial Infarction (MI)
  * No Prior Coronary Revascularization Procedures
  * No Patients with ≥ 70% Obstructive Coronary Disease

Exclusion Criteria:

* ST Elevation Myocardial Infarction (STEMI) Activation
* ST Changes or new T-wave inversions ≥1mm on ECG
* Any Elevated Troponin Measure (Based on Sex-Specific 99th Percentile)
* Serial change between Troponin Measures (Delta) ≥5 pg/mL
* Stress Echocardiography, Nuclear Stress Test, Stress ECG, Stress Cardiac MRI, Coronary CT Angiogram (CCTA), Invasive Coronary Angiography (Cardiac Cath) within 1 year
* "Clean" CCTA or Cardiac Cath (0% stenosis in all vessels) within the past 2 years
* Chest Trauma
* Pregnancy
* Life Expectancy < 1 year
* Other comorbid conditions requiring hospitalization
* Unstable Vitals (Blood Pressure <90, Heart Rate >120 or <50, O2 Sat <90%)
* End Stage Renal Disease; Dialysis or estimated glomerular filtration rate (eGFR) <30 mL/min
* Transfers From Another Hospital
* Non-English Speaking
* Prisoners
* Prior Enrollment
* Already Enrolled in Other Interventional Trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Hospital-free days (HFD) at 30-days post-randomization | Day 30
  Time spent in a hospital setting at 30 days post-randomization will be measured and subtracted from time spent outside the hospital. Hospital time is broadly defined, based on a patient-centered definition of cumulative time spent in the ED, observation unit, or hospital ward. Consistent with prior trials, patients who experience death during the follow-up period are assigned zero HFDs.

SECONDARY OUTCOMES:
Hospital-free days (HFD) at 1-year post-randomization | Year 1
  Time spent in a hospital setting at 1 year post-randomization will be measured and subtracted from time spent outside the hospital. Hospital time is broadly defined, based on a patient-centered definition of cumulative time spent in the ED, observation unit, or hospital ward. Consistent with prior trials, patients who experience death during the follow-up period are assigned zero HFDs.
Cardiovascular Hospital-free days (HFD) at 30-days post-randomization | Day 30
  Rates of cardiovascular rehospitalizations at 30-days post-randomization will be analyzed between the two treatment arms.
Cardiovascular Hospital-free days (HFD) at 1 year post-randomization | Year 1
  Rates of cardiovascular rehospitalizations at 1 year post-randomization will be analyzed between the two treatment arms.
Rate of noninvasive cardiac testing at 30-days post-randomization | Day 30
  The rates of noninvasive testing (stress testing and coronary computed tomography angiography), at 30-days post-randomization will be analyzed between the two treatment arms.
Rate of noninvasive cardiac testing at 1 year post-randomization | Year 1
  The rates of noninvasive testing (stress testing and coronary computed tomography angiography), at 1 year post-randomization will be analyzed between the two treatment arms.
Rate of invasive cardiac testing at 30-days post-randomization | Day 30
  The rates of invasive testing (coronary angiography), at 30-days post-randomization will be analyzed between the two treatment arms.
Rate of invasive cardiac testing at 1 year post-randomization | Year 1
  The rates of invasive testing (coronary angiography), at 1 year post-randomization will be analyzed between the two treatment arms.
Cardiovascular repeat ED visits at 30-days post-randomization | Day 30
  The rates of Cardiovascular repeat ED visits at 30-days post-randomization will be analyzed between the two treatment arms.The ED visit will be categorized as cardiovascular if a cardiac procedure is performed, the primary reason for admission is possible ACS, or a discharge diagnosis relates to chest pain, MI, ACS, heart failure, or other cardiac disease (e.g., dysrhythmia, pericardial disease, etc.). Cardiac procedures include stress testing, noninvasive and invasive coronary angiography, coronary revascularization, and pacemaker or defibrillator insertion.
Cardiovascular repeat ED visits at 1 year post-randomization | Year 1
  The rates of Cardiovascular repeat ED visits at 1 year post-randomization will be analyzed between the two treatment arms.The ED visit will be categorized as cardiovascular if a cardiac procedure is performed, the primary reason for admission is possible ACS, or a discharge diagnosis relates to chest pain, MI, ACS, heart failure, or other cardiac disease (e.g., dysrhythmia, pericardial disease, etc.). Cardiac procedures include stress testing, noninvasive and invasive coronary angiography, coronary revascularization, and pacemaker or defibrillator insertion.
Cardiovascular rehospitalizations at 30-days post-randomization | Day 30
  The rates of Cardiovascular rehospitalizations at 30-days post-randomization will be analyzed between the two treatment arms.The rehospitalization will be categorized as cardiovascular if a cardiac procedure is performed, the primary reason for admission is possible ACS, or a discharge diagnosis relates to chest pain, MI, ACS, heart failure, or other cardiac disease (e.g., dysrhythmia, pericardial disease, etc.). Cardiac procedures include stress testing, noninvasive and invasive coronary angiography, coronary revascularization, and pacemaker or defibrillator insertion.
Cardiovascular rehospitalizations at 1 year post-randomization | Year 1
  The rates of Cardiovascular rehospitalizations at 1 year post-randomization will be analyzed between the two treatment arms.The rehospitalization will be categorized as cardiovascular if a cardiac procedure is performed, the primary reason for admission is possible ACS, or a discharge diagnosis relates to chest pain, MI, ACS, heart failure, or other cardiac disease (e.g., dysrhythmia, pericardial disease, etc.). Cardiac procedures include stress testing, noninvasive and invasive coronary angiography, coronary revascularization, and pacemaker or defibrillator insertion.
Patient satisfaction (SAPS questionnaire) | Day 30
  Satisfaction will be assessed using the Short Assessment of Patient Satisfaction (SAPS). A patient satisfaction survey will be sent that evaluates clinician communication, participation in medical decision-making, respect by the clinician, clinician carefulness, time with the clinician, and treatment effect, in any service setting on a five-point Likert scale from "very dissatisfied" to "very satisfied". Scores from each item are summed and range from 0 (extremely dissatisfied) to 28 (extremely satisfied).
Patient experience (GS-PEQ instrument) | Day 30
  Experience will be measured using the Generic Short Patient Experience Questionnaire (GS-PEQ). A patient experience survey will also be sent out to evaluate which assesses timeliness and organization of medical services, confidence in the clinician and treatment, patient involvement in decision-making, clinician communication, patient outcomes, and incorrect treatment on a 5-point Likert-scale from "not at all" to "to a very large extent" and one question (on wait times) scored on a 4-point Likert scale from "no" to "yes, way too long. A mean score can be calculated for each patient, with higher scores indicating better experience.
Out-of-pocket cost (based on billing data) | Day 30
  Patient satisfaction, patient experience, and out-of-pocket costs will be measured in all trial participants. Financial records will be utilized from each site to determine patient billing, including the amount covered by insurance vs. patient responsibility. Each item will be measured in U.S. dollars and summed for total cost.
Drivers of Patient Satisfaction and Experience (Qualitative) | Day 30
  A subset of 100 patients (50 from each arm) will be purposively selected to ensure diversity in sex, race, ethnicity, socioeconomic status (SES), and health literacy for 30-minute semi-structured phone interviews to determine key drivers of patient satisfaction and experience. We will use an explanatory sequential mixed-methods design, in which participants' quantitative data will guide the collection and analysis of their qualitative data.These data will provide key context and meaning to the patient's quantitative response regarding patient satisfaction, experience, and out-of-pocket cost.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Mahler, MD, MS, Principal Investigator — Wake Forest University Health Sciences
Locations (3):
- United States (3):
  - Henry Ford Hospital, Detroit, Michigan
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No